CLINICAL TRIAL: NCT01247311
Title: The Impact of Vitamin D Supplementation on Vascular Stiffness and Blood Pressure in Chronic Kidney Disease Patients
Brief Title: Vitamin D and the Health of Blood Vessels in Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Kidney Foundation of Canada (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H10-01689
Record Dates: First submitted 2010-11-12; First posted 2010-11-24 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Vitamin D; pulse wave velocity
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dietary Supplements; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. (Active Comparator): 1,25 Vitamin D (0.50ug *3 per week)
  This is a prospective randomized double blind placebo controlled study of 125 stable CKD subjects examining the impact of vitamin D supplementation (1,25 vitamin D or 25 vitamin D formulations) compared to placebo on arterial stiffness and other parameters of vascular health
  Interventions: Dietary Supplement: Vitamin D
- 2. (Active Comparator): 25 Vitamin D (5000IU * 3 per week)
  This is a prospective randomized double blind placebo controlled study of 125 stable CKD subjects examining the impact of vitamin D supplementation (1,25 vitamin D or 25 vitamin D formulations) compared to placebo on arterial stiffness and other parameters of vascular health
  Interventions: Dietary Supplement: Vitamin D
- 3. (Placebo Comparator): Placebo given orally 3xweek for six months
  Interventions: Dietary Supplement: Dietary supplement

INTERVENTIONS:
Dietary Supplement: Dietary supplement — Placebo given orally 3xweek for six months
  Arms: 3.
Dietary Supplement: Vitamin D — 5000 IU vitamin D given orally 3xweek for six months
  Arms: 2.
Dietary Supplement: Vitamin D — 0.5ug 1,25 vitamin D given orally 3xweek for six months
  Arms: 1.

SUMMARY:
Individuals with kidney disease have a high risk of heart disease. This is not related to traditional risk factors, such as high blood pressure, high cholesterol or being overweight. A lack of vitamin D could be the reason why blood vessels become damaged and could explain the link between heart disease and kidney disease.

DETAILED DESCRIPTION:
Most people living in Canada do not receive enough vitamin D from the sun or from the food they eat. When a person has kidney disease this is a particular problem as kidney disease stops what little vitamin D we do have being activated in the body. Low levels of activated vitamin D causes a domino effect with calcium and phosphate and all the hormones that control calcium and phosphate. Some people believe that this imbalance damages the blood vessels causing them to become stiff and inflexible (arterial stiffness) and this in turn could cause heart disease. In addition there are two different types of vitamin D that can be prescribed and it is currently not known whether there is any difference between the two types of vitamin D and the effect they have on the blood vessels.

The purpose of this study is to investigate whether providing vitamin D as a medication can have a direct affect on the stiffness of the blood vessels. The findings of this study will help both physicians and dietitians decide whether Vitamin D therapy is beneficial to patients and should help decide which type of Vitamin D is best to give to people with chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* patients with an estimated glomerular filtration rate (eGFR) between 15 - 45 ml/min, and <2ml/min change in glomerular filtration rate (GFR) over the past 6 months
* treated with maximal conventional cardiovascular disease (CVD) risk reduction medications

Exclusion Criteria:

* patients with estimated glomerular filtration rate (eGFR) change of >2.1 ml/min over the past 6 months
* those who have terminal malignancies
* those with planned transplant within 6 months, or who are likely to commence renal replacement therapy (dialysis) within the 6 months after enrolment
* those with active infections or active inflammatory diseases (Systemic Lupus Erythematosus (SLE), vasculitis)
* those who refuse to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Help both physicians and dietitians decide whether vitamin D therapy is beneficial to patients with kidney disease | 15 months
  The specific measurements to establish the primary outcome measure include:a pulse wave velocity test which is a non-invasive test used to measure the elasticity of the blood vessels (randomized groups will be compared from baseline to 6 months); blood pressure measurements (randomized groups will be compared for rate of change in BP over 6 months); blood and urine collection (randomized groups will be compared for rate of change in proteinuria, fibroblast growth factor-23, serum parathyroid hormone, phosphate, calcium and C-reactive protein).

CONTACTS AND LOCATIONS:
Overall Officials: Adeera Levin, Dr., Principal Investigator — University of British Columbia
Locations (1):
- St Paul's Hospital & Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Levin A, Perry T, De Zoysa P, Sigrist MK, Humphries K, Tang M, Djurdjev O. A randomized control trial to assess the impact of vitamin D supplementation compared to placebo on vascular stiffness in chronic kidney disease patients. BMC Cardiovasc Disord. 2014 Nov 7;14:156. doi: 10.1186/1471-2261-14-156. PMID 25381032
- [Result] Levin A, Tang M, Perry T, Zalunardo N, Beaulieu M, Dubland JA, Zerr K, Djurdjev O. Randomized Controlled Trial for the Effect of Vitamin D Supplementation on Vascular Stiffness in CKD. Clin J Am Soc Nephrol. 2017 Sep 7;12(9):1447-1460. doi: 10.2215/CJN.10791016. Epub 2017 May 26. PMID 28550081